CLINICAL TRIAL: NCT02533570
Title: A Multi-center, Randomized, Double-blinded, Placebo-controlled, Multiple-ascending-dose Study of Brentuximab Vedotin in Adults With Active Systemic Lupus Erythematosus
Brief Title: Dose Ranging Study of Brentuximab Vedotin in Adults With Lupus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision based on portfolio prioritization
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SGN35-022
Record Dates: First submitted 2015-07-09; First posted 2015-08-27 (Estimated); Results first posted 2018-06-11 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-05

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Lupus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Brentuximab Vedotin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brentuximab vedotin (Experimental): 4 dose groups
  Interventions: Drug: Brentuximab vedotin
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Brentuximab vedotin
  Other Names: ADCETRIS (brentuximab vedotin)
  Arms: Brentuximab vedotin
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of brentuximab vedotin in adults with active systemic lupus erythematosus (SLE).

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a chronic, multisystem, disabling autoimmune condition, which predominantly affects women of childbearing years. Treatment options for SLE remain relatively limited. Regardless of the specific therapy chosen, the majority of patients continue to require long term immunomodulatory or cytotoxic therapy, resulting in long-term morbidity and mortality. Brentuximab vedotin is an antibody-drug conjugate (ADC) consisting of: 1) the chimeric immunoglobulin (Ig) G1 antibody cAC10, specific for human CD30, 2) the microtubule disrupting agent monomethyl auristatin E (MMAE), and 3) a protease-cleavable linker that covalently attaches MMAE to cAC10. Since CD30 and/or CD30-expressing immune cells may play significant key roles in the pathogenesis of SLE, brentuximab vedotin may be an efficacious therapy. This study intends to explore the potential for brentuximab vedotin as a therapy for SLE.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years
* Diagnosis of SLE for at least 6 months prior to screening
* Active SLE as indicated by SLE Disease Activity Index (SLEDAI) ≥ 4 at screening
* Must have failed a treatment for SLE after a trial of at least 3 months

Exclusion Criteria:

* The subject has any serious health condition, which, in the opinion of the Investigator, would place the subject at undue risk from the study
* Subject has had recent serious or ongoing infection, or risk for serious infection
* Subject has a history of new or recurrent malignancy within the past 5 years
* The subject is pregnant and/or breastfeeding
* The subject fulfills diagnostic criteria for another rheumatic (overlap) disease that may confound clinical assessments in the study
* The subject has urgent, severe SLE disease activity, which, in the opinion of the Investigator, warrants immediate immunosuppressive therapy and would not be appropriate for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-07; Primary Completion 2017-06-05 (Actual); Study Completion 2017-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Sesterhenn, MD, Study Director — Seattle Genetics Medical Monitor
Locations (17):
- United States (17):
  - University of Alabama at Birmingham - (UAB), Birmingham, Alabama
  - TriWest Research Associates, LLC, El Cajon, California
  - Advanced Medical Research, LLC, La Palma, California
  - University of Colorado, Aurora, Colorado
  - Clinical Research of West Florida - Corporate, Clearwater, Florida
  - Lakes Research, LLC, Miami Lakes, Florida
  - Arthritis Associates, Orlando, Florida
  - McIlwain Medical Group, Tampa, Florida
  - Henry Ford Health System, Detroit, Michigan
  - Clayton Medical Associates, P.C., St Louis, Missouri
  - Weill Cornell Physicians at Brooklyn Heights, Brooklyn, New York
  - DJL Clinical Research, PLLC, Charlotte, North Carolina
  - Arthritis & Rheumatology Center of Oklahoma, Oklahoma City, Oklahoma
  - Ramesh C Gupta MD, Memphis, Tennessee
  - Tekton Research, Inc., Austin, Texas
  - Accurate Clinical Research, Houston, Texas
  - Arthritis Clinic of Northern Virginia, PC, Arlington, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Intravenous (IV) placebo every 3 weeks for a total of 4 doses
- Brentuximab Vedotin 0.3 mg/kg: Intravenous (IV) Brentuximab vedotin (0.3 mg/kg) every 3 weeks for a total of 4 doses
- Brentuximab Vedotin 0.6 mg/kg: Intravenous (IV) Brentuximab vedotin (0.6 mg/kg) every 3 weeks for a total of 4 doses
Period: Overall Study
Arm/Group | Placebo | Brentuximab Vedotin 0.3 mg/kg | Brentuximab Vedotin 0.6 mg/kg
Started | 4 | 8 | 8
Completed | 4 | 7 | 7
Not Completed | 0 | 1 | 1
Not completed — Adverse Event | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Brentuximab Vedotin 0.3 mg/kg | Brentuximab Vedotin 0.6 mg/kg | Total
Number analyzed (Participants) | 4 | 8 | 8 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (8.66) | 50.8 (14.06) | 45.0 (11.20) | 47.4 (11.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 8 | 20
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 3 | 4
  Not Hispanic or Latino | 3 | 8 | 5 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 5 | 7
  White | 3 | 6 | 3 | 12
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 8 | 8 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Subjects Having an Adverse Event (AE)
Description: Any treatment-emergent adverse events (TEAEs), any drug-related TEAEs, any SAEs, treatment-related serious adverse events (SAE), deaths, adverse events (AEs) leading to study discontinuation, and number of patients experiencing Grade 1, 2, and 3 TEAEs.
Time Frame: Up to 127 days (9 weeks after final dose)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Brentuximab Vedotin 0.3 mg/kg | Brentuximab Vedotin 0.6 mg/kg
Number analyzed (Participants) | 4 | 8 | 8
Participants
  Treatment-Emergent Adverse Event | 3 | 6 | 8
  Treatment-Related Adverse Event | 0 | 3 | 1
  Serious Adverse Event | 0 | 1 | 1
  Treatment-Related Serious Adverse Events | 0 | 1 | 0
  Deaths | 0 | 0 | 0
  Adverse Events Leading to Study Discontinuation | 0 | 1 | 1
  Any Grade 1 Adverse Event | 2 | 6 | 2
  Any Grade 2 Adverse Event | 2 | 4 | 7
  Any Grade 3 Adverse Event | 0 | 1 | 2

2. Secondary Outcome: Proportion of Subjects Achieving an SRI Response at Day 85
Description: Assessment for response was made using data only for the visit of interest (Day 85), without regard for changes at prior on-treatment visits.
  SRI: SLE Responder Index; SLE: Systemic lupus erythematosus
Time Frame: 85 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Brentuximab Vedotin 0.3 mg/kg | Brentuximab Vedotin 0.6 mg/kg
Number analyzed (Participants) | 4 | 7 | 7
Participants | 0 | 1 | 2

ADVERSE EVENTS:
Time Frame: Up to 127 days (9 weeks after last dose). The safety reporting period for all AEs and SAEs is from the date of consent through the follow-up visit. All SAEs that occur after the safety reporting period and are considered study treatment-related in the opinion of the Investigator should also be reported to the Sponsor. Additionally, new-onset neuropathy, suspected PML, or other AEs/SAEs of interest are reported until the end of the follow-up period.
Arm/Group | Placebo | Brentuximab Vedotin 0.3 mg/kg | Brentuximab Vedotin 0.6 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/8 | 1/8
Other Adverse Events (participants affected / at risk) | 3/4 | 6/8 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=4) | Brentuximab Vedotin 0.3 mg/kg (N=8) | Brentuximab Vedotin 0.6 mg/kg (N=8)
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=4) | Brentuximab Vedotin 0.3 mg/kg (N=8) | Brentuximab Vedotin 0.6 mg/kg (N=8)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Infusion Site Pain (General disorders) | 0 | 1 | 0
Infusion Site Pruritus (General disorders) | 0 | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 1 | 0
Oedema Peripheral (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1
Fungal Infection (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0
Tinea Manum (Infections and infestations) | 0 | 0 | 1
Tinea Pedis (Infections and infestations) | 0 | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1
Avulsion Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tooth Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Limb Discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 3 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0
Mental Status Changes (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Ovarian Cyst (Reproductive system and breast disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermal Cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Vascular Compression (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The sponsor may extend the embargo for a period up to 60 days to allow for the filing of a one or more patent applications. The sponsor cannot require changes to the communication and cannot otherwise extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2016-07-25): https://cdn.clinicaltrials.gov/large-docs/70/NCT02533570/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-31): https://cdn.clinicaltrials.gov/large-docs/70/NCT02533570/SAP_001.pdf